CLINICAL TRIAL: NCT03803137
Title: Volatil Organic Compounds in Exhaled Air and Sweat After Thoracic Surgery for Carcinological Resection
Acronym: Onco-VOC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2017081
Record Dates: First submitted 2018-10-05; First posted 2019-01-14 (Actual); Last update posted 2020-12-19 (Actual); Status verified 2020-12

CONDITIONS: Lung Cancer, Non-small Cell
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VOC analysis (Experimental): VOC analysis in exhaled air and sweat in patients with thoracic surgery for carcinological resection
  Interventions: Other: VOC analysis

INTERVENTIONS:
Other: VOC analysis — VOC analysis in exhaled air with e-noses and mass spectrometry

SUMMARY:
Bronchopulmonary cancer, with 39 000 new cases and 30 000 deaths per year, is a main issue in public health in France. It is the leading cause of cancer death in France. A lot of progress in medical care has been made, but surgery remains the most effective treatment, when it is still possible. The goal is to detect and manage the lung cancer as early as possible. Alongside screening strategies by annual thoracic scanner, new approaches with innovative technologies open up for cancer detection and therapeutic follow-up.

The study of volatile organic compounds (VOC) detected in exhaled air or in sweat, is an innovative research area for respiratory diseases. The volatolomic analysis can be done either by the technique of the mass spectrometry which allows the identification of each VOC in the exhaled air or by the technique of electronic nose, simpler and faster, which provides an idea of the general profile of the VOC without identifying them. The VOC have shown their interest in some situations, such as diagnostic or prognostic tool in patients followed for thoracic tumorous pathology or bronchial or pulmonary vascular diseases.

The composition of VOC in exhaled air and sweat is altered in patients with lung cancer. The VOC analysis and their variation could be used particularly in the follow-up of patients treated for lung cancer.

The purpose of this clinical research is to identify the VOCs related to lung cancers by comparing the VOC profiles in exhaled air and in sweat from patients diagnosed with localized lung cancer before and after resection surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged ≥ 18 years old
* Patient with non-small cell lung cancer
* Operable grade I or II
* No specific treatment before surgery (radiotherapy, chemotherapy or targeted therapy)
* Patient with healthcare insurance

Non Inclusion Criteria:

* Treatment with radiotherapy, chemotherapy, or neoadjuvant cancer targeted therapy before thoracic surgery
* Patient with oxygen therapy or invasive ventilation
* Patient unable to perform a slow vital capacity
* Dermatological therapy interfering with sweat collection (psoriasis, irritant dermatitis, for instance)
* Pregnant women
* Patient deprived of liberty by judicial or administrative decision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-09-20 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Comparison of Volatil Organic Compound (VOC) profiles by mass spectrometry | change from baseline profiles at 2 month post-surgery
  Comparison of variation in Volatil Organic Compound (VOC) profiles in exhaled air of patients before and after surgery. The VOC will be identified by their molecular mass (by the mass spectrometry)
Comparison of Volatil Organic Compound (VOC) profiles in by electronic noses | change from baseline profiles at 2 month post-surgery
  Comparison of variation in Volatil Organic Compound (VOC) profiles in exhaled air of patients before and after surgery. The VOC will be identified by the sensor deflection (by the electronic noses).

SECONDARY OUTCOMES:
Comparison of Volatil Organic Compound (VOC) profiles in sweat | 30 days before the surgery and 45 to 75 days after surgery
  Comparison of Volatil Organic Compound (VOC) profiles in sweat of patients before and after surgery. The VOC will be identified by their molecular mass (by the mass spectrometry).
Variation of Volatil Organic Compound (VOC) and relapse rate | 30 days before the surgery, 45 to 75 days after surgery and 2 years
  Correlation between the variation of Volatil Organic Compound (VOC) before-after surgery and relapse rate at 2 years
Correlation between Volatil Organic Compound (VOC) profiles and relapse rate | 2 months and 2 years after surgery
  Correlation between the Volatil Organic Compound (VOC) profiles 2 months after the surgery and relapse rate at 2 years
Comparison of Volatil Organic Compound (VOC) profiles in exhaled air and tumoral lung tissue | 30 days before the surgery, day of surgery and 45 to 75 days after surgery
  Comparison of Volatil Organic Compound (VOC) profiles in exhaled air of patients and those released ex-vivo by the tumoral lung tissue. The VOC will be identified by their molecular mass (by the mass spectrometry).

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Devillier, Principal Investigator — Pneumology department
Locations (1):
- Hôpital Foch, Suresnes, France

IPD SHARING:
Plan to Share IPD: Undecided